CLINICAL TRIAL: NCT02782351
Title: Humanized CAR-T Therapy for Treatment of Recurrent or Refractory B Cell Malignancy by Targeting CD19
Brief Title: Humanized CAR-T Therapy for Treatment of B Cell Malignancy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kai Lin Xu; Jun Nian Zheng (Other)
Collaborators: iCarTAB BioMed Inc. (Unknown); Huaian first people's hospital (Unknown)
Responsible Party: Sponsor-Investigator, Kai Lin Xu; Jun Nian Zheng, President, Xuzhou Medical University
Organization: Xuzhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2016-KL002-01
Record Dates: First submitted 2016-05-17; First posted 2016-05-25 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CAR-T (Experimental): In interventional studies, patients enrolled will receive autologous 2nd generation CAR-T cells, which contain a humanized single chain antibody sequence against CD19.
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — Patients will be infused with autologous CAR-T infusion in a dose escalating manner.

SUMMARY:
The present study evaluates the safety and efficacy of humanized Chimeric antigen receptor T cells (CAR-T) in treating recurrent or refractory B cell malignancy targeting CD19 with a humanized scFv. All participants will receive autologous chimeric antigen receptor engineered T cells.

DETAILED DESCRIPTION:
CD19 has been extensively evaluated as a therapeutic target for recurrent or refractory B cell malignancy by chimeric antigen receptor T cell therapy, the single chain antibody sequence (scFv) against CD19 derived from a mouse hybridoma was widely employed. However, the immunogenicity of the mouse scFv sequence might be one of the reasons that CAR-T cells cannot persist in vivo for long. In present study investigators replace the mouse-derived scFv with a a humanized one and evaluate its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age≥3 at the time of consent
* Survival time>12 weeks
* B cell hematological malignancies by pathological examination
* Chemotherapy failure or recurrent B cell malignancy
* Creatinine< 2.5mg/dl
* Glutamic-pyruvic transaminase, glutamic oxalacetic transaminase< 3 fold of normal level
* Karnofsky Performance Status>50% at the time of screening
* Bilirubin<2.0mg/dl
* Adequate pulmonary, renal, hepatic, and cardiac function
* Fail in autologous or allogenic haemopoietic stem cell transplantation
* Free of leukocytes removal contraindications

Exclusion Criteria:

* Pregnant or nursing women
* Active hepatitis B, active hepatitis C, or any human immunodeficiency virus (HIV) infection at the time of screening
* Previous treatment with any gene therapy product
* Abnormal vital signs
* Highly allergic constitution or history of severe allergies, especially allergy to interleukin-2
* General infection or local severe infection, or other infection that is not controlled
* Dysfunction in lung, heart, kidney and brain.
* Severe autoimmune diseases
* other symptoms that are not applicable for CAR-T

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
CAR-T cells persistence in peripheral blood | 12 months
  The presence of CAR T cells in patients' peripheral blood will be quantified with real time qPCR

SECONDARY OUTCOMES:
B cell number and immunoglobulins in peripheral blood | 12 months
  The number of B cells and immunoglobulins in peripheral blood will be evaluated by routine methods

CONTACTS AND LOCATIONS:
Overall Officials: KaiLin Xu, MD. Ph.D., Principal Investigator — Xuzhou Medical University
Locations (2):
- China (2):
  - Huaian First People's Hospital, Huai'an, Jiangsu
  - Affiliated hospital of Xuzhou medical college, Xuzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] van der Stegen SJ, Hamieh M, Sadelain M. The pharmacology of second-generation chimeric antigen receptors. Nat Rev Drug Discov. 2015 Jul;14(7):499-509. doi: 10.1038/nrd4597. PMID 26129802
- [Result] Davila ML, Bouhassira DC, Park JH, Curran KJ, Smith EL, Pegram HJ, Brentjens R. Chimeric antigen receptors for the adoptive T cell therapy of hematologic malignancies. Int J Hematol. 2014 Apr;99(4):361-71. doi: 10.1007/s12185-013-1479-5. Epub 2013 Dec 6. PMID 24311149
- [Derived] Qi Y, Zhao M, Hu Y, Wang Y, Li P, Cao J, Shi M, Tan J, Zhang M, Xiao X, Xia J, Ma S, Qiao J, Yan Z, Li H, Pan B, Sang W, Li D, Li Z, Zhou J, Huang H, Liang A, Zheng J, Xu K. Efficacy and safety of CD19-specific CAR T cell-based therapy in B-cell acute lymphoblastic leukemia patients with CNSL. Blood. 2022 Jun 9;139(23):3376-3386. doi: 10.1182/blood.2021013733. PMID 35338773
- [Derived] Chen W, Ma Y, Shen Z, Chen H, Ma R, Yan D, Shi M, Wang X, Song X, Sun C, Cao J, Cheng H, Zhu F, Sun H, Li D, Li Z, Zheng J, Xu K, Sang W. Humanized Anti-CD19 CAR-T Cell Therapy and Sequential Allogeneic Hematopoietic Stem Cell Transplantation Achieved Long-Term Survival in Refractory and Relapsed B Lymphocytic Leukemia: A Retrospective Study of CAR-T Cell Therapy. Front Immunol. 2021 Oct 29;12:755549. doi: 10.3389/fimmu.2021.755549. eCollection 2021. PMID 34777367